CLINICAL TRIAL: NCT07179731
Title: Comparison of the Effects of External Oblique Intercostal Plane Block, Subcostal Transverse Abdominis Plane Block, and Their Combination in the Management of Postoperative Pain in Laparoscopic Cholecystectomy Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Faruk Komez, MD, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EOİKB001
Record Dates: First submitted 2025-07-31; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-07

CONDITIONS: External Oblique Intercostal Plane Block; Subcostal Transverse Abdominis Plane Block
Keywords: external oblique intercostal block; subcostal transverse abdominis block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: subcostal transversus abdominis plane block (Active Comparator): This group will receive 30 ml 0.25% of bupivacaine for the subcostal transversus abdominis plane block prior to surgery.
  Interventions: Procedure: subcostal transversus abdominis plane block
- Group 2: external oblique intercostal plane block (Active Comparator): This group will receive 30 ml 0.25% of bupivacaine for the external oblique intercostal plane block prior to surgery.
  Interventions: Procedure: External Oblique Intercostal Plane Block
- Group 3: subcostal transversus abdominis and external oblique intercostal plane block combination (Active Comparator): This group will receive 15 ml 0.25% of bupivacaine for the external oblique intercostal plane block, in combination with 15 ml 0.25% of bupivacaine for the subcostal transversus abdominis plane block prior to surgery.
  Interventions: Procedure: external oblique intercostal plane block and subcostal transversus abdominis plane block combination

INTERVENTIONS:
Procedure: subcostal transversus abdominis plane block — Under ultrasound guidance, 30 ml of bupivacaine is injected along the fascia of transversus abdominis muscle.
  Arms: Group 1: subcostal transversus abdominis plane block
Procedure: External Oblique Intercostal Plane Block — Under ultrasound guidance, 30 ml of bupivacaine is injected between the fascias of external oblique and intercostal muscles.
  Arms: Group 2: external oblique intercostal plane block
Procedure: external oblique intercostal plane block and subcostal transversus abdominis plane block combination — The combination of the two blocks will be applied in 15 ml of volume for each.
  Arms: Group 3: subcostal transversus abdominis and external oblique intercostal plane block combination

SUMMARY:
This study aims to compare the efficacy of Subcostal Transversus Abdominis Plan Block, External Oblique Intercostal Plan Block and the combination of these two blocks, which are used in anesthesiology practice for postoperative pain in laparoscopy cholecystectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laparoscopic cholecystectomy surgery
* Patients aged between 18 to 80 years
* Having an anesthesiology risk assessment of ASA I, II, or III

Exclusion Criteria:

* Patients who do not give written and oral consent
* Patients with coagulopathy
* History of allergic reaction or intoxication by local anesthetics
* Severe organ failure
* Mental retardation or illiteracy
* Presence of infection on the injection site
* Pregnancy
* Patients whom the procedure is extended to open cholecystectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-09-23 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Analgesic Consumption | 24 hours postoperatively
  The opioid consumption via patient controlled analgesia (PCA) in 24 hours postoperatively

SECONDARY OUTCOMES:
Postoperative Pain Scores | up to 24 hours after surgery
  Postoperative pain will be assessed using Numeric Rating Scale (NRS) at 30 mins, and 1, 4, 8, 12, 24 hours after surgery.

IPD SHARING:
Plan to Share IPD: No